CLINICAL TRIAL: NCT03935568
Title: A Single and Multiple Ascending Dose Study to Evaluate the Safety and Pharmacokinetics of PU-AD in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company ceased operations
Sponsor: Samus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PU-AD-01-001
Record Dates: First submitted 2019-04-24; First posted 2019-05-02 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Alzheimer's Disease
Keywords: PU-AD
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Single Dose Placebo (Experimental): Patients randomized to receive Placebo
  Interventions: Drug: Placebo
- Single Dose Active (PU-AD) (Experimental): Patients randomized to receive Active (PU-AD)
  Interventions: Drug: PU-AD
- Multiple Dose (Placebo) (Experimental): Patients randomized to receive Placebo
  Interventions: Drug: Placebo
- Multiple Dose Active (PU-AD) (Experimental): Patients randomized to receive Active (PU-AD)
  Interventions: Drug: PU-AD

INTERVENTIONS:
Drug: PU-AD — 3 cohorts receiving a single oral dose of PU-AD at one time.
  Arms: Single Dose Active (PU-AD)
Drug: Placebo — 3 cohorts receiving a single oral dose of Placebo at one time
  Arms: Single Dose Placebo
Drug: Placebo — 2 cohorts receiving multiple oral dose of Placebo at one time
  Arms: Multiple Dose (Placebo)
Drug: PU-AD — 2 cohorts receiving multiple oral dose of PU-AD at one time
  Arms: Multiple Dose Active (PU-AD)

SUMMARY:
This is a first in human Phase 1 study in two parts with healthy volunteers receiving a single dose of PU AD in three small cohorts and a multiple ascending dose in two small cohorts.

DETAILED DESCRIPTION:
This is a Phase 1, double-blind trial in two parts. A single ascending dose study in approximately 3 cohorts receiving a single oral dose of PU-AD or placebo and a multiple ascending dose study in 2 cohorts. Each subject in all cohorts will be administered an oral solution of PU AD or placebo under fasting conditions. Each cohort will contain subjects randomized to active treatment or placebo, evaluating safety and tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (Women of non-child bearing potential)
2. 18 to 60 years of age for part one, >/= 60 years of age for part two

Exclusion Criteria:

1. Women of child bearing potential or Female with positive pregnancy test or who is lactating.
2. History or presence of conditions, which in the judgment of the PI, are known to interfere with the absorption distribution, metabolism, or excretion of drugs.
3. History or presence of conditions that may place the subject at increased risk as determined by the PI.
4. Has taken other investigational drugs or participated in any clinical study within 30 days.
5. Any other condition or prior therapy that, in the PI's opinion, would make the subject unsuitable for the study, or unable or unwilling to comply with the study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple doses of PU-AD in healthy subjects | Day 1 to Day 3
  Adverse Event (AE) incidence and changes from baseline in clinical laboratory test results. Number and percentage of subjects reporting any treatment emergent AE will be tabulated by system organ class and preferred term for each treatment (coded using Medical Dictionary for Regulatory Activities). Treatment-emergent AEs will be further classified by severity and relationship to treatment.
To evaluate the safety and tolerability of single and multiple doses of PU-AD in healthy subjects | Day 1 to Day 3
  Adverse event incidence and changes from baseline in Electrocardiogram. Number and percentage of subjects reporting any treatment emergent AE will be tabulated by system organ class and preferred term for each treatment (coded using Medical Dictionary for Regulatory Activities). Treatment-emergent AEs will be further classified by severity and relationship to treatment.
To evaluate the safety and tolerability of single and multiple doses of PU-AD in healthy subjects | Day 1 to Day 3
  Adverse event incidence and changes from baseline in vital signs . Number and percentage of subjects reporting any treatment emergent AE will be tabulated by system organ class and preferred term for each treatment (coded using Medical Dictionary for Regulatory Activities). Treatment-emergent AEs will be further classified by severity and relationship to treatment.

SECONDARY OUTCOMES:
To determine the pharmacokinetics (PK) PU-AD in healthy subjects | Day 1 to Day 3
  Collect PK parameters to estimate human exposure,after dose administration for each cohort will be evaluated using a power model for dose proportionality. (Maximum observed concentration (Cmax).
To determine the pharmacokinetics (PK) PU-AD in healthy subjects | Day 1 to Day 3
  Collect PK parameters to estimate human exposure,after dose administration for each cohort will be evaluated using a power model for dose proportionality. (Time to maximum observed concentration (tmax).
To determine the pharmacokinetics (PK) PU-AD in healthy subjects | Day 1 to Day 3
  Collect PK parameters to estimate human exposure,after dose administration for each cohort will be evaluated using a power model for dose proportionality. (Area under the concentration-time curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, M.D., Study Director — Samus Therapeutics
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silverman MH, Duggan S, Bardelli G, Sadler B, Key C, Medlock M, Reynolds L, Wallner B. Safety, Tolerability and Pharmacokinetics of Icapamespib, a Selective Epichaperome Inhibitor, in Healthy Adults. J Prev Alzheimers Dis. 2022;9(4):635-645. doi: 10.14283/jpad.2022.71. PMID 36281667